CLINICAL TRIAL: NCT06785532
Title: Investigating the Effect of Responsive Neurostimulation (RNS) in Patients with Treatment-refractory Tourette's Syndrome (TR-TS)
Brief Title: Effect of RNS in Treatment-refractory Tourette's Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNS for TRTS
Record Dates: First submitted 2025-01-14; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Tourette Syndrome
Keywords: TS, RNS
MeSH Terms: conditions — Tourette Syndrome; Raine syndrome

STUDY DESIGN:
Intervention Model Description: Patients with Treatment-refractory Tourette's syndrome (TR-TS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment-refractory Tourette's Syndrome (TR-TS) (Experimental): Patients will undergo bilateral RNS lead implantation.
  Interventions: Device: Responsive Neurostimulation (RNS)

INTERVENTIONS:
Device: Responsive Neurostimulation (RNS) — The RNS lead is stereotactically introduced into the target in the brain and fixed to the skull; the lead is then connected to a neurostimulator implanted subcutaneously in the subclavicular region.

SUMMARY:
The study is to investigate the effect of personalized responsive neurostimulation (RNS) therapy guided by stereoelectroencephalography (SEEG) in patients with treatment-resistant Tourette's Syndrome (TR-TS).

DETAILED DESCRIPTION:
Tourette's Syndrome (TS) is a neurodevelopmental disorder characterized by repetitive, involuntary movements and vocalizations known as tics. It typically manifests in childhood and may persist into adulthood. The prevalence of TS varies globally, affecting approximately 1% of the population. There is a broad spectrum of symptom severity. Treatment-refractory TS (TR-TS) refers to cases where standard therapeutic interventions, such as behavioural therapy and medications, have shown limited effectiveness. TR-TS prevalence is relatively lower but highlights the challenges in managing severe and persistent symptoms. In a comprehensive survey of diverse neuromodulation therapies, targeting specific nuclei with personalized responsive neurostimulation (RNS) has the most potential for TR-TS with apparent symptoms. However, the RNS case reports are limited and lack high-quality, evidence-based medical evidence. The stimulation targets of RNS for patients with TS include GPi, amGPi, pvGPi, Cm-Spv-Voi, Cm-Voi, and NA-ALIC. While stereoelectroencephalography (SEEG) brain mapping can help identify Individualized effective targets and stimulation parameters. So, this cohort study focuses on the effectiveness of SEEG-guided RNS on TR-TS patients. Another goal is to study the neuronal activity of the GPi, amGPi, pvGPi, Cm-Spv-Voi, Cm-Voi, and NA-ALIC, or other unreported nuclei targets, respectively. At the same time, some subjects are presented with a task involving an unexpected reward and different cognitive tasks.

Some participants will also be invited to join a related study that involves positron emission tomography (PET) scanning to determine how the stimulation changes activity in the brain. Participation in the separate PET study is optional.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65;
2. able to provide written informed consent;
3. have a diagnosis of Tourette's syndrome according to the Statistical Manual of Mental Disorders-Fourth Edition-Text Revised (DSM-IV-TR) criteria and confirmed by the Mini-International Neuropsychiatric Interview Chinese version 5.0;
4. with a YGTSS of at least 35 for at least 12 months before surgery, while YGTSS- Total Motor≥15;
5. must have failed conventional medical treatment at adequate therapeutic doses of three classes of medication lasting for at least three months;
6. must not be suitable for behavioural intervention or that this intervention is inappropriate or unsuccessful;
7. have been on stable comorbid conditions without suicidal ideation for at least six months.

Exclusion Criteria:

1. presence of other psychotic disorders;
2. have a treatment history that includes electroconvulsive therapy (ECT), modified electroconvulsive therapy (MECT), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), DBS, and transcranial magnetic stimulation (TMS);
3. presents a suicide risk (defined as a HAMD-17 score of ≥3 on suicide-related items);
4. experience difficulty in effectively communicating with investigators;
5. with a history of traumatic brain injury (TBI);
6. with intracranial or cardiovascular stents;
7. substance abuse within the past six months;
8. unstable neurological or coagulation disorders;
9. women who are pregnant, lactating, or of childbearing potential who refuse the use of reliable contraception during the study;
10. have been involved in other clinical studies within three months before enrollment in this study;
11. any conditions considered by the study group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS): Reduction in total tics on the YGTSS after 12 months | Baseline to 12 months post-surgery
  The YGTSS is a 10-item semi-structured clinician-rating instrument that evaluates motor and phonic symptoms' number, frequency, intensity, complexity, and interference. The items about the tic ratings are scored on two subscales: motor tics and phonic tics. Behaviors are rated on a 6-point scale. The Total Tic Severity Score ranges from 0-50, with a higher score indicating a higher severity of symptoms.

SECONDARY OUTCOMES:
YGTSS-Total Motor: Change in YGTSS-Total Motor at week 2, month 3, month 6, and month 12. | Baseline to week 2, month 3, month 6, and month 12
  The YGTSS motor tics are rated on a 6-point scale. The score ranges from 0-25, with a higher score indicating a higher severity of symptoms.
YGTSS-Total Phonic: Change in YGTSS-Total phonic at week 2, month 3, month 6, and month 12. | Baseline to week 2, month 3, month 6, and month 12
  The YGTSS phonic tics are rated on a 6-point scale. The score ranges from 0-25, with a higher score indicating a higher severity of symptoms.
YGTSS: remission. | Baseline to week 2, month 3, month 6, and month 12
  Remission (defined as YGTSS total score ≤14) at Week 2, Month 3, Month 6, and Month 12.
YGTSS: response rate. | Baseline to week 2, month 3, month 6, and month 12
  Response is a ≥35% reduction in YGTSS total score from baseline to Week 2, Month 3, Month 6, and Month 12.
Yale-Brown Obsessive Compulsive Scale (Y-BOCS): Change in Y-BOCS at week 2, month 3, month 6, and month 12. | Baseline to week 2, month 3, month 6, and month 12
  The Y-BOCS scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms), yielding a total possible score range from 0 to 40. The total score is usually computed from the subscales for obsessions (items 1-5) and compulsions (items 6-10). The results can be interpreted based on the total score: 0-7 is sub-clinical; 8-15 is mild; 16-23 is moderate; 24-31 is severe; 32-40 is extreme. The Y-BOCS scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms), yielding a total possible score range from 0 to 40. The total score is usually computed from the subscales for obsessions (items 1-5) and compulsions (items 6-10). The results can be interpreted based on the total score: 0-7 is sub-clinical; 8-15 is mild; 16-23 is moderate; 24-31 is severe; 32-40 is extreme.
Hamilton Anxiety Scale (HAMA): the change from baseline to 2 weeks, 3 months, 6 months, and 12 months in the HAMA total score. | Baseline to week 2, month 3, month 6, and month 12
  HAMA is a 14-item test measuring the severity of anxiety symptoms. The total anxiety score ranges from zero to 56, with higher scores indicating more anxiety. The seven psychic anxiety items elicit a psychic anxiety score that ranges from 0 to 28. The remaining seven items yield a somatic anxiety score ranging from 0 to 28.
Hamilton Depression Rating Scale (HAMD-17): the changes of HAMD-17 scores and its subscales from baseline to 2 weeks, 3 months, 6 months, and 12 months. | Baseline to week 2, month 3, month 6, and month 12
  Hamilton Depression Rating Scale (HAMD-17): the changes of HAMD-17 scores and its subscales from baseline to 2 weeks, 3 months, 6 months, and 12 months.
Pittsburgh Sleep Quality Index (PSQI): the change of PSQI from baseline to Week 2, Month 3, Month 6, and Month 12. | Baseline to week 2, month 3, month 6, and month 12
  Consisting of 19 items, the PSQI measures several aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Clinical Global Impression-Severity (CGI-S): the change from baseline to 2 weeks, 3 months, 6 months, and 12 months in Clinical Global Impression-Severity (CGI-S) Remove | Baseline to week 2, month 3, month 6, and month 12
  The clinical global impression-severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. Score 1 presents normal, not at all ill, and score 7 presents among the most extremely ill patients.
Clinical Global Impression-Improvement (CGI-I): CGI-I score at Week 2, Month 1, Month 3, Month 6, and Month 12. | Baseline to week 2, month 3, month 6, and month 12
  The clinical global impression-improvement scale (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Score 1 presents the patient as much improved, and score 7 presents much worse.
EuroQol-5 Dimension-level Scale (EQ-5D-5L): the change from baseline to Week 2, Month 3, Month 6, and Month 12 in EQ-5D-5L. | Baseline to week 2, month 3, month 6, and month 12
  EQ-5D-5L is an instrument that evaluates the generic quality of life. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The score ranges from 5 (having no problems) to 25 (being unable to do/having extreme problems).
Young Mania Rating Scale (YMRS): the change from baseline to Week 2, Month 1, Month 3, Month 6, and Month 12. | Baseline to week 2, month 3, month 6, and month 12
  This scale has 11 items and is based on the patient's subjective report of his or her clinical condition over the previous 48 hours. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Scores range from 0 to 60, with higher scores indicating more severe mania. A score of 0 to 5 means no obvious manic symptoms; a score of 6 to 10 means definite manic symptoms; a score of 22 or above means severe manic symptoms. It will be used as a systematic screen for DBS-induced mania or hypomania. Although scores above 8 have been considered evidence of manic symptomatology in bipolar patients, the unmasked physician will use this scale and screening questions to assess whether any hypomanic symptoms require clinical intervention including DBS adjustment.
Safety as indicated by the number of Adverse Events: Week 2, Month 3, Month 6, and Month 12. | Baseline to week 2, month 3, month 6, and month 12
  Possible Adverse Events include: Major and minor adverse events will be evaluated by Adverse Events Questionnaire (AEQ) and accompanying Case Report Form (AEQ CRF) in multiple domains, including psychiatric, neurological, and cognitive effects. The AEQ includes cognitive and behavioral screening items used in the Xuanwu DBS clinic for movement disorder patients. Additionally, we have added items for the adverse events observed in pilot DBS for TR-TS.
Change from baseline in the Verbal Fluency Test (COWAT) | 1 year after neurostimulator implantation.
  During the Controlled Oral Word Association Test (COWAT), individuals are tasked with verbally generating words starting with different letters of the alphabet. They have 60 seconds for each letter to retrieve and articulate as many words as possible. The test involves presenting three letters, each progressively more challenging in associative difficulty. Scores are derived by summing the total words produced across the three letter trials. The lowest achievable score is zero, indicating an inability to generate any words. There is no upper limit to the score as participants can produce numerous words for each letter. Higher scores reflect superior word retrieval and cognitive function.
Change from baseline in the Trailmaking Test A&B | 1 year after neurostimulator implantation.
  The Trail Making Test A and B assess cognitive shifting, visual search speed, scanning, processing speed, mental flexibility, and executive functioning. It evaluates the participant's capacity for sequencing (Parts A and B), cognitive set shifting (Part B), and processing speed (Parts A and B). Scores for Part A and Part B are calculated independently, indicating the number of seconds required for the participant to finish each section. Higher scores denote longer durations for completing the test.
Change in Rey-Osterrieth Complex Figure Test | 1 year after neurostimulator implantation.
  The Rey-Osterrieth complex figure test (ROCF) is a neuropsychological assessment in which patients are asked to reproduce a complicated line drawing, first by copying it freehand (recognition), and then drawing from memory (recall). Scoring of drawings is based on the widely used 36-point scoring system (0 being the worst score and 36 the best).

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Wang, MD & PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided